CLINICAL TRIAL: NCT06304922
Title: BRCA 1/2 Status as a Predictive Factor to Response to Platinum Based Chemotherapy in Cancer Ovary
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nesreen Haidra Ahmed Garad, Principal investigator, Assiut University
Other Study IDs: BRCA 1/2 in cancer ovary
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Assess the response to platinum-based chemotherapy in correlation to BRCA status in neoadjuvant and recurrent ovarian cancer — Assess the response to platinum-based chemotherapy in correlation to BRCA status in neoadjuvant and recurrent ovarian cancer

SUMMARY:
The main objective of this prospective study is to assess the clinical outcomes of platinum based chemotherapy cases either cisplatin or carboplatin according to BRCA status in neoadjuvant and recurrent ovarian cancer.

DETAILED DESCRIPTION:
Ovarian cancer was the third most common gynecological cancer globally in 2020. Ovarian carcinoma is the most common type of ovarian cancer, comprising over 90% of all ovarian cancer cases.

It is the most lethal gynecologic malignancy in high-income countries.

Approximately, 10-15% of epithelial ovarian cancer (EOC) patients carry germline mutation in BRCA1 or BRCA2. But,the majority of cases are sporadic.

Increased body mass index (BMI) and hormone replacement therapy (HRT) have been proposed as major contributors along with smoking and occupational hazards e.g., asbestos exposure.

Studies have reported that the prevalence of BRCA mutations varies among different epithelial ovarian ca ( EOC) subtypes, with prevalence of 20%-25% reported for the high-grade serous subtype , BRCA mutations were reported in <10% of the endometrioid subtype and with very low frequency in clear cell subtype (6.3%).

The absence of BRCA1/2 function is associated with a cumulative lifetime risk for developing epithelial ovarian cancer of 40% to 50% in patients who are BRCA1-mutation carriers and 20% to 25% in patients who are BRCA2-mutation carriers.

Improved prognosis in terms of progression-free survival (PFS) and overall survival (OS), with higher partial response (PR) and complete response (CR) rates to platinum-containing regimens and longer treatment-free intervals, has been observed in retrospective studies of patients who are BRCA1/2-mutant carriers with ovarian cancer compared with patients who are non.

However, despite a generally favorable response to first-line chemotherapy, the disease frequently recurs. Due to limited therapeutic options, sequential chemotherapy regimens are often used based on platinum sensitivity (determined by the platinum-free interval), residual toxicities, general condition/performance status, and co-morbidities, with suboptimal outcomes and cumulative toxicity. Treatment effectiveness decreases over time, with resistance to platinum drugs precluding diminished survival and quality of life.

Germ-line BRCA mutations are associated with longer survival rates after ovarian cancer diagnosis and generally favorable response to platin-based therapy.

No data available for recurrent cases to assess the response of platinum based chemotherapy in BRCA mutant or wild cases.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years,
* Pathologically proven ovarian cancer,epithelial origin.
* BRCA mutant/wild
* Recurrent cases who are eligible to anti-VEGF (Bevacizumab).
* Patients with clinical stages T1-T3c , N0-N1b, M0, and recurrent platinum sensitive cases.
* Patients with good renal and liver functions.
* No other malignancy (double malignancy).
* Performance status 0-2 according to ECOG performance status scale.

Exclusion Criteria:

* Performance status 3-4 according to ECOG performance status scale.
* Patients refuse to receive chemotherapy,
* Patients not eligible to receive chemotherapy due to liver or renal impairment.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Ovarian cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate. | 1 year
  percentage of people in the study or treatment group who have a partial response or complete response to the treatment within a certain period of time; wil be correlated with BRCA status.
Progression free survival | 1 year
  the time from starting the study till disease progression or death from any cause

SECONDARY OUTCOMES:
Overall survival and toxicity | 2 years
  the length of time from either the date of diagnosis or start of treatment for cancer ovary are still alive

REFERENCES:
- [Background] Huang J, Chan WC, Ngai CH, Lok V, Zhang L, Lucero-Prisno DE 3rd, Xu W, Zheng ZJ, Elcarte E, Withers M, Wong MCS, On Behalf Of Ncd Global Health Research Group Of Association Of Pacific Rim Universities Apru. Worldwide Burden, Risk Factors, and Temporal Trends of Ovarian Cancer: A Global Study. Cancers (Basel). 2022 Apr 29;14(9):2230. doi: 10.3390/cancers14092230. PMID 35565359
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Manchana T, Phoolcharoen N, Tantbirojn P. BRCA mutation in high grade epithelial ovarian cancers. Gynecol Oncol Rep. 2019 Aug 13;29:102-105. doi: 10.1016/j.gore.2019.07.007. eCollection 2019 Aug. PMID 31467961
- [Background] Whelan E, Kalliala I, Semertzidou A, Raglan O, Bowden S, Kechagias K, Markozannes G, Cividini S, McNeish I, Marchesi J, MacIntyre D, Bennett P, Tsilidis K, Kyrgiou M. Risk Factors for Ovarian Cancer: An Umbrella Review of the Literature. Cancers (Basel). 2022 May 30;14(11):2708. doi: 10.3390/cancers14112708. PMID 35681688
- [Background] Brown KF, Rumgay H, Dunlop C, Ryan M, Quartly F, Cox A, Deas A, Elliss-Brookes L, Gavin A, Hounsome L, Huws D, Ormiston-Smith N, Shelton J, White C, Parkin DM. The fraction of cancer attributable to modifiable risk factors in England, Wales, Scotland, Northern Ireland, and the United Kingdom in 2015. Br J Cancer. 2018 Apr;118(8):1130-1141. doi: 10.1038/s41416-018-0029-6. Epub 2018 Mar 23. PMID 29567982
- [Background] Liu H, Zhang Z, Chen L, Pang J, Wu H, Liang Z. Next-Generation Sequencing Reveals a Very Low Prevalence of Deleterious Mutations of Homologous Recombination Repair Genes and Homologous Recombination Deficiency in Ovarian Clear Cell Carcinoma. Front Oncol. 2022 Jan 12;11:798173. doi: 10.3389/fonc.2021.798173. eCollection 2021. PMID 35096598
- [Background] Jazaeri AA. Molecular profiles of hereditary epithelial ovarian cancers and their implications for the biology of this disease. Mol Oncol. 2009 Apr;3(2):151-6. doi: 10.1016/j.molonc.2009.01.001. Epub 2009 Feb 7. PMID 19383376
- [Background] Coburn SB, Bray F, Sherman ME, Trabert B. International patterns and trends in ovarian cancer incidence, overall and by histologic subtype. Int J Cancer. 2017 Jun 1;140(11):2451-2460. doi: 10.1002/ijc.30676. Epub 2017 Mar 21. PMID 28257597
- [Background] Pujade-Lauraine E, Banerjee S, Pignata S. Management of Platinum-Resistant, Relapsed Epithelial Ovarian Cancer and New Drug Perspectives. J Clin Oncol. 2019 Sep 20;37(27):2437-2448. doi: 10.1200/JCO.19.00194. Epub 2019 Aug 12. No abstract available. PMID 31403868
- [Background] Alsop K, Fereday S, Meldrum C, deFazio A, Emmanuel C, George J, Dobrovic A, Birrer MJ, Webb PM, Stewart C, Friedlander M, Fox S, Bowtell D, Mitchell G. BRCA mutation frequency and patterns of treatment response in BRCA mutation-positive women with ovarian cancer: a report from the Australian Ovarian Cancer Study Group. J Clin Oncol. 2012 Jul 20;30(21):2654-63. doi: 10.1200/JCO.2011.39.8545. Epub 2012 Jun 18. PMID 22711857
- [Background] Tan DS, Kaye SB. Chemotherapy for Patients with BRCA1 and BRCA2-Mutated Ovarian Cancer: Same or Different? Am Soc Clin Oncol Educ Book. 2015:114-21. doi: 10.14694/EdBook_AM.2015.35.114. PMID 25993149